CLINICAL TRIAL: NCT04148937
Title: A Phase 1 Multicenter Global First in Human Study of the CD73 Inhibitor LY3475070 as Monotherapy or in Combination With Pembrolizumab in Patients With Advanced Solid Malignancies
Brief Title: A Study of the CD73 Inhibitor LY3475070 Alone or in Combination With Pembrolizumab in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17504; J2I-MC-JZMA (Other: Eli Lilly and Company); 2019-003270-64 (EudraCT Number); Keynote A57 (Other: Merck)
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cancer
Keywords: Triple Negative Breast Cancer; Pancreatic Cancer; Non-small Cell Lung Cancer; Renal Cell Carcinoma, Clear Cell; Cutaneous Melanoma; Castrate Resistant Prostate Cancer; Epithelial Ovarian Cancer; Metastatic Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Carcinoma, Ovarian Epithelial; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1a Cohort A LY3475070 (dose escalation) (Experimental): Participants received 150 milligram (mg) once daily or 300 mg once daily or 300mg twice daily or 600mg once daily oral LY3475070 on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
  Interventions: Drug: LY3475070
- Phase 1a Cohort B LY3475070 + Pembrolizumab (dose escalation) (Experimental): Participants received 150 mg once daily or 150 mg twice daily or 300 mg once daily or 300mg twice daily oral LY3475070 on a 21-day cycle in combination with an intravenous infusion of 200mg pembrolizumab on day 1 until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
  Interventions: Drug: LY3475070; Drug: Pembrolizumab
- Phase 1b Cohort C1 LY3475070 + Pembrolizumab (dose expansion) (Experimental): LY3475070 administered orally and pembrolizumab administered IV.
  Based on Sponsor decision, Phase 1b expansion cohorts were not initiated.
  Interventions: Drug: LY3475070; Drug: Pembrolizumab
- Phase 1b Cohort C2 LY3475070 (dose expansion) (Experimental): LY3475070 administered orally.
  Based on Sponsor decision, Phase 1b expansion cohorts were not initiated.
  Interventions: Drug: LY3475070
- Phase 1b Cohort D1 LY3475070 + Pembrolizumab (dose expansion) (Experimental): LY3475070 administered orally and pembrolizumab administered IV.
  Based on Sponsor decision, Phase 1b expansion cohorts were not initiated.
  Interventions: Drug: LY3475070; Drug: Pembrolizumab
- Phase 1b Cohort D2 LY3475070 (dose expansion) (Experimental): LY3475070 administered orally.
  Based on Sponsor decision, Phase 1b expansion cohorts were not initiated.
  Interventions: Drug: LY3475070
- Phase 1b Cohort E LY3475070 + Pembrolizumab (dose expansion) (Experimental): LY3475070 administered orally and pembrolizumab administered IV.
  Based on Sponsor decision, Phase 1b expansion cohorts were not initiated.
  Interventions: Drug: LY3475070; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LY3475070 — Administered orally
Drug: Pembrolizumab — Administered IV
  Arms: Phase 1a Cohort B LY3475070 + Pembrolizumab (dose escalation); Phase 1b Cohort C1 LY3475070 + Pembrolizumab (dose expansion); Phase 1b Cohort D1 LY3475070 + Pembrolizumab (dose expansion); Phase 1b Cohort E LY3475070 + Pembrolizumab (dose expansion)

SUMMARY:
The reason for this study is to see if the CD73 inhibitor LY3475070 alone or in combination with pembrolizumab is safe and effective in participants with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have certain types of cancer such as breast cancer, pancreatic cancer, lung cancer, kidney cancer, skin cancer (melanoma), prostate cancer, and ovarian cancer
* Participants must have stopped other forms of treatment for the cancer
* In the expansion cohorts participants must be able and willing to provide a sample of the tumor before beginning treatment and a sample during the treatment. For certain tumor types, the result of a test on the tumor sample may exclude the participant from the study
* Participants must not be pregnant, and must agree to use birth control
* Participants must have progressed through or be intolerant to therapies with known clinical benefit

Exclusion Criteria:

* Participants must not have a current untreated tuberculosis, lung disease, heart disease, uncontrolled HIV, autoimmune disease, active hepatitis B or C virus infection or using corticosteroids
* Participant must not have cancer that has spread to the brain
* Participant must not have received a vaccine within the last 30 days
* Participant must not have had bowel obstruction within the last 6 months, or intestinal surgery
* Participant must not have an infection that is currently being treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (7):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists ORLANDO/DDU, Lake Mary, Florida
  - START Midwest, Grand Rapids, Michigan
  - Washington University Medical School, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Beatson West of Scotland Cancer Center, Glasgow, Scotland
  - Christie NHS Foundation Trust, Manchester
  - Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of the CD73 Inhibitor LY3475070 Alone or in Combination With Pembrolizumab in Participants With Advanced Cancer — https://trials.lillytrialguide.com/en-US/trial/3IgVmdVs6HVWj9kMys9jsd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially designed to be conducted in two phases: Phase 1a (dose escalation cohorts A, B) and Phase 1b (dose expansion cohorts C1, C2, D1, D2, E). Based on Sponsor decision, Phase 1b expansion cohorts were not initiated, no participants were enrolled.
Groups:
- Cohort A - 150mg QD LY3475070: Participants received 150 milligrams (mg) LY3475070 orally once daily (QD) on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort A - 300mg QD LY3475070: Participants received 300mg LY3475070 orally once daily on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort A - 300mg BID LY3475070: Participants received 300mg LY3475070 orally twice daily (BID) on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort A - 600mg QD LY3475070: Participants received 600mg LY3475070 orally once daily on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort B - 150mg QD LY3475070 + Pembrolizumab: Participants received 150mg LY3475070 orally once daily on a 21-day cycle in combination with an intravenous infusion of 200mg pembrolizumab on day 1 until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort B - 150mg BID LY3475070 + Pembrolizumab: Participants received 150mg LY3475070 orally twice daily on a 21-day cycle in combination with an intravenous infusion of 200mg pembrolizumab on day 1 until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort B - 300mg QD LY3475070 + Pembrolizumab: Participants received 300mg LY3475070 orally once daily on a 21-day cycle in combination with an intravenous infusion of 200mg pembrolizumab on day 1 until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort B - 300mg BID LY3475070 + Pembrolizumab: Participants received 300mg LY3475070 orally twice daily on a 21-day cycle in combination with an intravenous infusion of 200mg pembrolizumab on day 1 until progressive disease, unacceptable toxicity or other criterion for study
Period: Overall Study
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Started | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Received at Least 1 Dose of Study Drug | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Completed (Completers include participants who were observed until event (progressive disease or death) or had discontinued study treatment and was in follow up at the time of the final analysis.) | 4 | 6 | 5 | 3 | 3 | 8 | 0 | 17
Not Completed | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab | Total
Number analyzed (Participants) | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.50 (9.57) | 65.83 (13.04) | 66.83 (12.22) | 66.25 (13.02) | 63.67 (7.23) | 59.73 (11.65) | 61 (0) | 66 (7.66) | 64.58 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 1 | 5 | 1 | 2 | 17
  Male | 2 | 3 | 4 | 3 | 2 | 6 | 0 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  White | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 14 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 6 | 3 | 2 | 8 | 1 | 13 | 38
  United Kingdom | 2 | 3 | 0 | 1 | 1 | 3 | 0 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as an adverse event that is likely related to the study medication or combination, and fulfils any one of the following criteria, graded according to the NCI-CTCAE (National Cancer Institute-Common Terminology Criteria for Adverse Events) version 5.0:
  * Grade 3 thrombocytopenia associated with clinically significant bleeding and requiring platelet transfusion or Grade 4 thrombocytopenia of any duration.
  * Grade ≥3 febrile neutropenia
  * Grade ≥3 anemia requiring a blood transfusion
  * Other Grade ≥4 toxicities, excluding few nonhematologic Toxicities
  * Any other significant toxicity deemed by the investigatory to be dose-limiting, such as: any toxicity that is possibly related to the study medication that requires the withdrawal of the participant from the study during 28-day DLT observation period), persistent Grade >2 toxicities causing a delay of LY3475070 study treatment >14 days during the 28-day DLT observation period.
Time Frame: Up to 28 days from the first dose
Population: All participants enrolled in the phase 1a who either completed 28 days of follow-up and at least 75% of LY3475070 treatment doses or discontinued treatment prior to 28 days due to a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A - 150mg QD LY3475070: Participants received 150mg LY3475070 orally once daily on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
- Cohort A - 300mg BID LY3475070: Participants received 300mg LY3475070 orally twice daily on a 21-day cycle until progressive disease, unacceptable toxicity or other criterion for study discontinuation is met.
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Eight Hours (AUC[0-8]) of LY3475070
Description: PK: AUC[0-8] of LY3475070.
Time Frame: Cycle 1 Day 1 (Pre-dose, 0.5, 1, 2, 4, 6, 8 hours post-dose)
Population: All enrolled participants in phase1a who received LY3475070 and had intensively sampled evaluable PK data on cycle 1 day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 5 | 4 | 3 | 7 | 1 | 13
nanograms*hours per milliliter (ng*h/mL) | 5880 (38.7) | 6580 (83.2) | 10700 (93.3) | 16000 (43.9) | 2990 (57.4) | 3680 (65.8) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 12600 ng*h/mL | 8960 (43.4)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve During 1 Dosing Interval (AUCtau) of LY3475070
Description: PK: AUCtau of LY3475070
Time Frame: Cycle 2 Day 1 (Pre-dose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose for the QD arms, Pre-dose, 0.5, 1, 2, 4, 6, 8 hours post-dose for the BID arms)
Population: All enrolled participants in phase1a who received LY3475070 and had intensively sampled evaluable PK data on cycle 2 day 1. For "Cohort B - 300mg QD LY3475070 + pembrolizumab," the participant has not received the treatment on cycle 2 day 1, and did not meet the analysis criteria. Thus, zero participants were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 3 | 3 | 3 | 6 | 0 | 12
ng*h/mL | 7950 (73.6) | 8320 (106) | 19600 (117) | 26200 (11.4) | 3180 (152) | 3280 (370) |  | 12400 (80.2)

4. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3475070
Description: PK: Cmax of LY3475070
Time Frame: Day 1 of Cycles 1 and 2 (Pre-dose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose for the QD arms; Pre-dose, 0.5, 1, 2, 4, 6, 8 hours post-dose for the BID arms)
Population: All enrolled participants in phase1a who received LY3475070 and had intensively sampled evaluable PK data on cycle 1 day 1, cycle 2 day 1 for this outcome. For "Cohort B - 300mg QD LY3475070 + pembrolizumab," the participant has not received the treatment on cycle 2 day 1, and did not meet the analysis criteria. Thus, zero participants were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 5 | 4 | 3 | 8 | 1 | 15
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 6 | 5 | 4 | 3 | 8 | 1 | 14
  Cycle 1 Day 1 | 1750 (13.2) | 2060 (61.3) | 2960 (113) | 4320 (29.2) | 1100 (63.1) | 974 (107) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there was only one participant. Individual value reported: 3270 ng/mL | 2670 (39.6)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 6 | 3 | 3 | 3 | 8 | 0 | 15
  Cycle 2 Day 1 | 1770 (32.9) | 2310 (105) | 4270 (87.5) | 4610 (17.2) | 1340 (72.2) | 1060 (170) |  | 3200 (58.2)

5. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: ORR is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline through Disease Progression or Death (Estimated at up to 10.4 Months)
Population: All enrolled participants in phase1a who received at least one dose of LY3475070.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and Stable Disease (SD)
Description: DCR is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Estimated at up to 10.4 Months)
Population: All enrolled participants in phase1a who received at least one dose of LY3475070.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Percentage of participants | 50 | 33.3 | 16.7 | 0 | 66.7 | 27.3 | 0 | 35.3

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of start of treatment to the first date of the observed clinical or radiologically documented progressive disease or death due to any cause, whichever occurs first, was estimated and reported for all evaluable participants. For participants who were not known to have died or progressed as of the data-inclusion cut-off date, PFS time was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Estimated at up to 10.4 Months)
Population: All enrolled participants in phase1a who received at least one dose of LY3475070 (including censored). Number of participants censored: 150mg QD LY3475070=1, 300mg QD LY3475070=1, 300mg BID LY3475070=4, 600mg QD LY3475070=1, 150mg QD LY3475070 + pembrolizumab=2, 150mg BID LY3475070 + pembrolizumab=5, 300mg QD LY3475070 + pembrolizumab=1, 300mg BID LY3475070 + pembrolizumab=14.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
Number analyzed (Participants) | 4 | 6 | 6 | 4 | 3 | 11 | 1 | 17
Months | 2.71 [0.03 to 3.42] | 1.91 [0.03 to 4.8] | 0.89 [0.03 to 2.14] | 1.33 [0.03 to 2.04] | 2 [0.03 to 2.04] | 0.53 [0.03 to 3.52] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 2.5]

ADVERSE EVENTS:
Time Frame: Baseline up to 10.4 months
Description: All enrolled participants in phase1a who received at least one dose of LY3475070. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Cohort A - 150mg QD LY3475070 | Cohort A - 300mg QD LY3475070 | Cohort A - 300mg BID LY3475070 | Cohort A - 600mg QD LY3475070 | Cohort B - 150mg QD LY3475070 + Pembrolizumab | Cohort B - 150mg BID LY3475070 + Pembrolizumab | Cohort B - 300mg QD LY3475070 + Pembrolizumab | Cohort B - 300mg BID LY3475070 + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 4/4 | 5/6 | 1/6 | 2/4 | 1/3 | 3/11 | 0/1 | 3/17
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 2/4 | 1/3 | 3/11 | 1/1 | 7/17
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 6/6 | 4/4 | 2/3 | 11/11 | 1/1 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - 150mg QD LY3475070 (N=4) | Cohort A - 300mg QD LY3475070 (N=6) | Cohort A - 300mg BID LY3475070 (N=6) | Cohort A - 600mg QD LY3475070 (N=4) | Cohort B - 150mg QD LY3475070 + Pembrolizumab (N=3) | Cohort B - 150mg BID LY3475070 + Pembrolizumab (N=11) | Cohort B - 300mg QD LY3475070 + Pembrolizumab (N=1) | Cohort B - 300mg BID LY3475070 + Pembrolizumab (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A - 150mg QD LY3475070 (N=4) | Cohort A - 300mg QD LY3475070 (N=6) | Cohort A - 300mg BID LY3475070 (N=6) | Cohort A - 600mg QD LY3475070 (N=4) | Cohort B - 150mg QD LY3475070 + Pembrolizumab (N=3) | Cohort B - 150mg BID LY3475070 + Pembrolizumab (N=11) | Cohort B - 300mg QD LY3475070 + Pembrolizumab (N=1) | Cohort B - 300mg BID LY3475070 + Pembrolizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 8 (10)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 4 (8)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (3) | 2 (3) | 3 (3) | 2 (5) | 0 (0) | 4 (4) | 1 (1) | 5 (10)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyp (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/2 (0) | 0/3 (0) | 1/2 (1) | 0/1 (0) | 0/1 (0) | 0/5 (0) | 0 (0) | 0/2 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (6)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tanning (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04148937/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04148937/SAP_001.pdf